CLINICAL TRIAL: NCT03295175
Title: Distribution of Smooth Muscle In Dartos In The Non Conspicuous Penis, an Observational a Prospective, Descriptive, Observational Study
Brief Title: Distribution of Smooth Muscle In Dartos In The Non Conspicuous Penis
Acronym: DISMUD
Status: Withdrawn | Type: Observational
Why Stopped: The project never started and contact with the main researcher was lost.
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Other Study IDs: FM-CIE-0319-17
Record Dates: First submitted 2017-09-24; First posted 2017-09-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Congenital Urogenital Anomaly
Keywords: Congenital Abnormalities; Hypospadias; Congenital megaprepuce; Histology
MeSH Terms: conditions — Urogenital Abnormalities; Congenital Abnormalities; Hypospadias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Congenital Megaprepuce: Congenital Megaprepuce Hematoxylin-eosin and smooth muscle actin markers
  Interventions: Diagnostic Test: Hematoxylin-eosin and smooth muscle actin markers
- Hypospadias: Hypospadias Hematoxylin-eosin and smooth muscle actin markers
  Interventions: Diagnostic Test: Hematoxylin-eosin and smooth muscle actin markers
- Control: Circumcision for non-medical reasons. Hematoxylin-eosin and smooth muscle actin markers
  Interventions: Diagnostic Test: Hematoxylin-eosin and smooth muscle actin markers

INTERVENTIONS:
Diagnostic Test: Hematoxylin-eosin and smooth muscle actin markers — The foreskin arrives oriented in a single piece in formol to the unit of pathology, and in the pathology unit, they must:
  1. Measure the length, width and thickness of the specimen. The specimen should include skin and mucosa with the underlying areolar tissue.
  2. Examine the surfaces of the sample searching lesions, and describe them in size, appearance (warty, papillary, ulcerated), depth of invasion, and distance from the nearest cutting edge, if they are present.

SUMMARY:
Non-conspicuous penis (congenital megaprepuce, occult penis) is a symptomatic malformation that includes phimosis and excessively baggy, urine-filled prepuce with alteration of the appearance of the penis. A redundant and enlarged foreskin is the main feature of this entity.This congenital anomaly is difficult to diagnose and may have association with other pathologies such as buried penis.

Currently, part of the megaprepuce skin is used to correct the defect. A recent study shows that patients with this pathology and hypospadias present mostly defects in the muscle dartos. The investigators do not know the physiological bases of the megaprepuce, neither the clinical and aesthetics implications of this abnormal tissue for the patient, and how this affects the postoperative evolution. With the present study the investigators intended to answer these questions and to open paths for future research in this area.

DETAILED DESCRIPTION:
After informed consent, patients will be labeled with a research record number other than the identity document or the number of the attention. The urologist who perform the correction of the megaprepuce, will take a segment of the dartos and send it for histopathological analysis: staining with hematoxylin-eosin, smooth muscle actin marker, associated with the research record number. Same procedure will be performed with the controls and hypospadias group. Only the principal investigator will know the assignment of medical record and their respective group (congenital megaprepuce, hypospadias or controls). The samples will be sent to pathology without any clinical data, and they will be analyzed by two pathologists, both blind.

ELIGIBILITY:
Inclusion Criteria:

* Male patients scheduled for correction of congenital megaprepuce
* Male patients scheduled for correction of hypospadias
* Male patients scheduled for circumcision for non-medical reasons.

Exclusion Criteria:

* Patients with a history of hypospadias correction.

Ages: 1 Month to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Male patients diagnosed with congenital megaprepuce and hypospadias scheduled for surgical correction.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Differences in the distribution of the smooth Muscle In Dartos | 1 year
  Smooth Muscle Fibers
Describe the pattern of smooth muscle in patients with megaprepuce | 1 year
  Smooth Muscle Fibers

SECONDARY OUTCOMES:
Describe the pattern of smooth muscle in patients with hypospadias | 1 year
  Smooth Muscle Fibers

CONTACTS AND LOCATIONS:
Overall Officials: Jose N Fernandez, MD, Principal Investigator — H
Locations (1):
- Luis Gabriel Villarraga, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruiz E, Vagni R, Apostolo C, Moldes J, Rodriguez H, Ormaechea M, Giuseppucci C, de Badiola F, Bortagaray J, Perea C. Simplified surgical approach to congenital megaprepuce: fixing, unfurling and tailoring revisited. J Urol. 2011 Jun;185(6 Suppl):2487-90. doi: 10.1016/j.juro.2011.01.015. Epub 2011 Apr 27. PMID 21527191
- [Result] Summerton DJ, McNally J, Denny AJ, Malone PS. Congenital megaprepuce: an emerging condition--how to recognize and treat it. BJU Int. 2000 Sep;86(4):519-22. doi: 10.1046/j.1464-410x.2000.00509.x. PMID 10971284
- [Result] Rod J, Desmonts A, Petit T, Ravasse P. Congenital megaprepuce: a 12-year experience (52 cases) of this specific form of buried penis. J Pediatr Urol. 2013 Dec;9(6 Pt A):784-8. doi: 10.1016/j.jpurol.2012.10.010. Epub 2012 Oct 30. PMID 23116700
- [Result] Alexander A, Lorenzo AJ, Salle JL, Rode H. The Ventral V-plasty: a simple procedure for the reconstruction of a congenital megaprepuce. J Pediatr Surg. 2010 Aug;45(8):1741-7. doi: 10.1016/j.jpedsurg.2010.03.033. PMID 20713233
- [Result] Borsellino A, Spagnoli A, Vallasciani S, Martini L, Ferro F. Surgical approach to concealed penis: technical refinements and outcome. Urology. 2007 Jun;69(6):1195-8. doi: 10.1016/j.urology.2007.01.065. PMID 17572214
- [Result] Spinoit AF, Van Praet C, Groen LA, Van Laecke E, Praet M, Hoebeke P. Congenital penile pathology is associated with abnormal development of the dartos muscle: a prospective study of primary penile surgery at a tertiary referral center. J Urol. 2015 May;193(5):1620-4. doi: 10.1016/j.juro.2014.10.090. Epub 2014 Oct 23. PMID 25444989
- [Result] Cimador M, Catalano P, Ortolano R, Giuffre M. The inconspicuous penis in children. Nat Rev Urol. 2015 Apr;12(4):205-15. doi: 10.1038/nrurol.2015.49. Epub 2015 Apr 7. PMID 25850928
- [Result] Maizels M, Zaontz M, Donovan J, Bushnick PN, Firlit CF. Surgical correction of the buried penis: description of a classification system and a technique to correct the disorder. J Urol. 1986 Jul;136(1 Pt 2):268-71. doi: 10.1016/s0022-5347(17)44837-3. PMID 2873259
- [Result] Crawford BS. Buried penis. Br J Plast Surg. 1977 Jan;30(1):96-9. doi: 10.1016/s0007-1226(77)90046-7. PMID 836989
- [Result] Shenoy MU, Rance CH. Surgical correction of congenital megaprepuce. Pediatr Surg Int. 1999;15(8):593-4. doi: 10.1007/s003830050683. PMID 10631746
- [Result] Hadidi AT. Buried penis: classification surgical approach. J Pediatr Surg. 2014 Feb;49(2):374-9. doi: 10.1016/j.jpedsurg.2013.09.066. Epub 2013 Nov 7. PMID 24528990
- [Result] Baskin LS, Himes K, Colborn T. Hypospadias and endocrine disruption: is there a connection? Environ Health Perspect. 2001 Nov;109(11):1175-83. doi: 10.1289/ehp.011091175. PMID 11713004
- [Result] Baskin LS, Ebbers MB. Hypospadias: anatomy, etiology, and technique. J Pediatr Surg. 2006 Mar;41(3):463-72. doi: 10.1016/j.jpedsurg.2005.11.059. PMID 16516617
- [Result] Fernandez N, Lorenzo A, Bagli D, Zarante I. Altitude as a risk factor for the development of hypospadias. Geographical cluster distribution analysis in South America. J Pediatr Urol. 2016 Oct;12(5):307.e1-307.e5. doi: 10.1016/j.jpurol.2016.03.015. Epub 2016 Apr 22. PMID 27267992